CLINICAL TRIAL: NCT03345823
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Maintenance and Long-Term Extension Study of the Efficacy and Safety of Upadacitinib (ABT-494) in Subjects With Crohn's Disease Who Completed the Studies M14-431 or M14-433
Brief Title: A Maintenance and Long-Term Extension Study of the Efficacy and Safety of Upadacitinib (ABT-494) in Participants With Crohn's Disease Who Completed the Studies M14-431 or M14-433
Acronym: U-ENDURE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-430; 2023-504951-29 (Other: EU CT)
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Crohn's Disease
Keywords: Upadacitinib; ABT-494; Extension Study; Efficacy; Safety; Crohn's Disease; Maintenance Study
MeSH Terms: conditions — Crohn Disease | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Substudy 1: Cohort 1 Upadacitinib Dose A (Experimental): This is a maintenance group which includes participants who achieved clinical response to upadacitinib in studies M14-431 and M14-433 and will receive upadacitinib dose A for 52 weeks.
  Interventions: Drug: Upadacitinib
- Substudy 1: Cohort 1 Upadacitinib Dose B (Experimental): This is a maintenance group which includes participants who achieved clinical response to upadacitinib in studies M14-431 and M14-433 and will receive upadacitinib dose B for 52 weeks.
  Interventions: Drug: Upadacitinib
- Substudy 1: Cohort 1 Placebo (Experimental): This is a maintenance group which includes participants who achieved clinical response to upadacitinib in studies M14-431 and M14-433 and will receive placebo for 52 weeks.
  Interventions: Drug: Placebo for Upadacitinib
- Substudy 1: Cohort 2 Placebo (Experimental): This is a maintenance group which includes participants who received double-blind placebo in studies M14-431 and M14-433 and achieved clinical response will continue to receive blinded placebo for 52 Weeks.
  Interventions: Drug: Placebo for Upadacitinib
- Substudy 1: Cohort 3 Upadacitinib Dose B (Experimental): This is a maintenance group which includes participants who achieved clinical response to upadacitinib from the extended treatment period of studies M14-431 and M14-433 and will receive upadacitinib Dose B for 52 Weeks.
  Interventions: Drug: Upadacitinib
- Substudy 2: Cohort 4 Upadacitinib Dose B (Experimental): This is a long-term extension group which includes participants who achieved clinical response in the open-label extended treatment period of study M14-431 and will receive upadacitinib dose B for 240 weeks.
  Interventions: Drug: Upadacitinib
- Substudy 2: Cohort 5 Upadacitinib Dose A (Experimental): This is a long-term extension group which includes participants who complete Substudy 1 and will receive upadacitinib dose A for 240 weeks.
  Interventions: Drug: Upadacitinib
- Substudy 2: Cohort 5 Upadacitinib Dose B (Experimental): This is a long-term extension group which includes participants who complete Substudy 1 and will receive upadacitinib dose B for 240 weeks.
  Interventions: Drug: Upadacitinib
- Substudy 2: Cohort 5 Placebo (Experimental): This is a long-term extension group which includes participants who complete Substudy 1 and will receive placebo for 240 weeks.
  Interventions: Drug: Placebo for Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — Oral; Tablet
  Other Names: ABT-494; RINVOQ
  Arms: Substudy 1: Cohort 1 Upadacitinib Dose A; Substudy 1: Cohort 1 Upadacitinib Dose B; Substudy 1: Cohort 3 Upadacitinib Dose B; Substudy 2: Cohort 4 Upadacitinib Dose B; Substudy 2: Cohort 5 Upadacitinib Dose A; Substudy 2: Cohort 5 Upadacitinib Dose B
Drug: Placebo for Upadacitinib — Oral; Tablet
  Arms: Substudy 1: Cohort 1 Placebo; Substudy 1: Cohort 2 Placebo; Substudy 2: Cohort 5 Placebo

SUMMARY:
A multicenter study to evaluate the efficacy and safety of maintenance and long-term treatment administration of upadacitinib, an orally administered Janus kinase 1 inhibitor, in adult participants with Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria:

For Substudy 1:

* Participant who achieve clinical response in Study M14-431 or Study M14-433.
* Participant completes study procedures in the parent study. The final endoscopy for Studies M14-431 or M14-433 may be missing, if the endoscopy cannot be performed during the COVID-19 pandemic.

For Substudy 2:

* Participant completes Substudy 1. The Week 52 endoscopy may be missing, if the endoscopy cannot be performed during the COVID-19 pandemic.
* Participant who achieved clinical response at the time described in the protocol and completes study procedures in the parent study/ substudy.

Exclusion Criteria:

For Substudies 1 and 2:

* Participant is considered by the investigator, for any reason, to be an unsuitable candidate for the study.
* Participant who has a known hypersensitivity to upadacitinib or its excipients, or had an adverse event during Studies M14-431 and M14-433 or Substudy 1 or 2 of Study M14-430 that in the investigator's judgment makes the participant unsuitable for this study.
* Participant at the final visit of M14-431 or M14-433 with any active or chronic recurring infections based on the investigator's assessment that makes the participant an unsuitable candidate for the study. Participants with serious infections undergoing treatment may be enrolled BUT NOT dosed until the infection treatment has been completed and the infection is resolved, based on the investigator's assessment.
* Participants with high grade colonic dysplasia or malignancy diagnosed at the endoscopy performed at the final visit of Studies M14-431, M14-433 or Substudy 1 of Study M14-430 (Week 52).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 747 (Estimated)
Dates: Start 2018-03-21 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Sub-Study 1: Percentage of Participants with Clinical Remission per Crohn's Disease Activity Index (CDAI) | Week 52
  Clinical remission per CDAI is defined as CDAI <150.
Sub-Study 1: Percentage of Participants with Endoscopic Response | Week 52
  Endoscopic response is defined as decrease in Simple Endoscopic Score for Crohn's Disease (SES-CD) from Baseline.
Number of Participants with Adverse Events | Through Week 240
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. For more details on adverse events please see the Adverse Event section.

SECONDARY OUTCOMES:
Sub-Study 1: Percentage of Participants with Clinical Remission per Patient-Reported Outcomes (PROs) | Week 52
  Clinical remission is defined based on average daily stool frequency (SF) AND average daily abdominal pain (AP) score.
Sub-Study 1: Percentage of Participants Achieving Clinical Response 100 (CR-100) | Week 52
  Decrease of at least 100 points in CDAI from Baseline.
Sub-Study 1: Percentage of Participants with Endoscopic Remission | Week 52
  Endoscopic remission is defined per Simplified Endoscopic Score for Crohn's Disease (SES-CD).
Sub-Study 1: Percentage of Participants without Corticosteroid use for Crohn's Disease Among All Participants | Week 52
  This is assessed in participants not taking corticosteroids at least 90 days prior to Week 52 and achieved clinical remission per CDAI. Clinical remission is defined as CDAI <150.
Sub-Study 1: Percentage of Participants with Clinical Remission per CDAI and Endoscopic Remission | Week 52
  Clinical remission per CDAI is defined as CDAI <150. Endoscopic remission is defined per SES-CD.
Sub-Study 1: Percentage of Participants with Clinical Remission per CDAI | Through Week 52
  Clinical remission per CDAI is defined as CDAI <150 (as measured by the percentage of participants with clinical remission at Week 52 among those with clinical remission at Week 0).
Sub-Study 1: Percentage of Participants who Discontinue Corticosteroid Use for Crohn's Disease at Least 90 Days Prior to Week 52 and Achieve Clinical Remission, in Participants Taking Corticosteroids at Baseline. | Week 52
  This is assessed in participants taking corticosteroids at Baseline. Clinical remission is defined based on average daily stool frequency (SF) AND average daily abdominal pain (AP) score.
Sub-Study 1: Change in Inflammatory Bowel Disease Questionnaire (IBDQ) | Baseline (Week 0) to Week 52
  The IBDQ is used to assess the quality of life of patients with inflammatory bowel disease.
Sub-Study 1: Change in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | Baseline (Week 0) to Week 52
  The FACIT-F questionnaire was developed to assess fatigue.
Sub-Study 1: Percentage of Participants with Hospitalizations due to Crohn's Disease (CD) | Up to Week 52
  This is assessed by reviewing participant's hospitalization data.
Sub-Study 1: Percentage of Participants with Resolution of Extra-Intestinal Manifestation (EIMs) , in Participants with EIMs at Baseline | Week 52
  EIMs are defined as manifestations of Crohn's disease in areas of the body other than the digestive tract, including eyes, skin, joints, mouth, and liver.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (466):
- United States (123):
  - East View Medical Research, LLC /ID# 171132, Mobile, Alabama
  - CB Flock Research Corporation /ID# 166239, Mobile, Alabama
  - Delsol Research Management, Ll /Id# 170164, Chandler, Arizona
  - Duplicate_HonorHealth Research Institute - Shea /ID# 164725, Scottsdale, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC /ID# 164702, Sun City, Arizona
  - Southern California Res. Ctr. /ID# 169653, Coronado, California
  - Citrus Valley Gastroenterology /ID# 166230, Covina, California
  - Hoag Memorial Hosp Presbyterian /ID# 222538, Irvine, California
  - UC San Diego Health System /ID# 164763, La Jolla, California
  - United Medical Doctors /ID# 207458, Los Alamitos, California
  - Gastrointestinal Biosciences Clinical Trials, LLC /ID# 164640, Los Angeles, California
  - Facey Medical Foundation /ID# 203138, Mission Hills, California
  - United Medical Doctors - Murrieta /ID# 164602, Murrieta, California
  - Medical Assoc Research Grp /ID# 169704, San Diego, California
  - UCSF Medical Center - Mount Zion /ID# 202372, San Francisco, California
  - Univ of California San Francis /ID# 164653, San Francisco, California
  - Care Access Research /ID# 167765, San Pablo, California
  - Peak Gastroenterology Associates, PC /ID# 170166, Colorado Springs, Colorado
  - Delta Waves, Inc. /ID# 164656, Colorado Springs, Colorado
  - Western States Clinical Res /ID# 164625, Wheat Ridge, Colorado
  - Gastroenterology Center of Connecticut /ID# 164614, Hamden, Connecticut
  - Advanced Research - Coral Springs /ID# 218019, Coral Springs, Florida
  - Encore Borland-Groover Clinical Research /Id# 203500, Jacksonville, Florida
  - Ctr for Advanced Gastroenterol /ID# 165306, Maitland, Florida
  - Crystal Pharmacology Research /ID# 166118, Miami, Florida
  - Coral Research Clinic /ID# 164604, Miami, Florida
  - Advanced Research Institute, Inc /ID# 164601, New Port Richey, Florida
  - Endoscopic Research, Inc. /ID# 206139, Orlando, Florida
  - Omega Research Group /ID# 203482, Orlando, Florida
  - Duplicate_Clinical Research of West Florida, Inc /ID# 205828, Tampa, Florida
  - Duplicate_Clinical Research of West Florida, Inc /ID# 208119, Tampa, Florida
  - Clinical Research Trials of Florida, Inc. /ID# 203486, Tampa, Florida
  - Duplicate_AdventHealth Tampa /ID# 171181, Tampa, Florida
  - Gastroenterology Associates of Central Georgia, LLC /ID# 165492, Macon, Georgia
  - Gastroenterology Consultants, P.C /ID# 218218, Roswell, Georgia
  - Atlanta Gastroenterology Spec /ID# 164698, Suwanee, Georgia
  - Treasure Valley Medical Research /ID# 215030, Boise, Idaho
  - Duplicate_Rush University Medical Center /ID# 165470, Chicago, Illinois
  - University of Chicago Medicine /ID# 165509, Chicago, Illinois
  - DuPage Medical Group /ID# 205320, Downers Grove, Illinois
  - MediSphere Medical Research Center /ID# 166233, Evansville, Indiana
  - Indianapolis Gastroenterology /ID# 164649, Indianapolis, Indiana
  - Aquiant Research /ID# 205505, New Albany, Indiana
  - University of Iowa Hospitals and Clinics /ID# 165405, Iowa City, Iowa
  - Tri-State Gastroenterology /ID# 165469, Crestview Hills, Kentucky
  - Duplicate_University of Louisville /ID# 165391, Louisville, Kentucky
  - University of Louisville Hospital /ID# 168520, Louisville, Kentucky
  - Houma Digestive Health Special /ID# 164727, Houma, Louisiana
  - Nola Research Works, LLC /ID# 164612, New Orleans, Louisiana
  - Louisiana Research Center, LLC /ID# 164694, Shreveport, Louisiana
  - Duplicate_Johns Hopkins University School of Medicine /ID# 211939, Baltimore, Maryland
  - Metropolitan Gastroenterology Group - Chevy Chase /ID# 164647, Chevy Chase, Maryland
  - Gastro Center of Maryland /ID# 171180, Columbia, Maryland
  - Duplicate_Lahey Hospital and Medical Center /ID# 214724, Burlington, Massachusetts
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 164654, Ann Arbor, Michigan
  - Clin Res Inst of Michigan, LLC /ID# 170163, Chesterfield, Michigan
  - Digestive Health Associates (DHA) - Farmington Hills /ID# 206101, Farmington Hills, Michigan
  - Center for Digestive Health /ID# 164726, Troy, Michigan
  - Mayo Clinic - Rochester /ID# 164691, Rochester, Minnesota
  - Southern Therapy and Advanced Research (STAR) LLC /ID# 165295, Jackson, Mississippi
  - Quality Clinical Research Inc. /ID# 170162, Omaha, Nebraska
  - CHI Health Research Center /ID# 168513, Omaha, Nebraska
  - Las Vegas Medical Research /ID# 168551, Las Vegas, Nevada
  - Cooper Gastroenterology at Fire Road /ID# 164641, Egg Harbor, New Jersey
  - Rutgers Robert Wood Johnson /ID# 166110, New Brunswick, New Jersey
  - NY Scientific /ID# 164630, Brooklyn, New York
  - United Health Services Hospitals, Inc /ID# 217483, Johnson City, New York
  - NYU Langone Long Island Clinical Research Associates /ID# 164627, Lake Success, New York
  - The Mount Sinai Hospital /ID# 170256, New York, New York
  - Columbia Univ Medical Center /ID# 164692, New York, New York
  - Gastoenterology Group of Rochester /ID# 166235, Rochester, New York
  - Richmond University Medical Center /ID# 201858, Staten Island, New York
  - Montefiore Medical Center - Moses Campus /ID# 166242, The Bronx, New York
  - Advantage Clinical Trials /ID# 168582, The Bronx, New York
  - Atrium Health Carolinas Medical Center /ID# 164632, Charlotte, North Carolina
  - Duplicate_PMG Research of Charlotte /ID# 171178, Charlotte, North Carolina
  - Wake Radiology UNC REX Healthcare - Raleigh Office /ID# 164752, Raleigh, North Carolina
  - Duplicate_Atrium Health Wake Forest Baptist Medical Center /ID# 164755, Winston-Salem, North Carolina
  - Plains Clinical Research Center, LLC /ID# 170169, Fargo, North Dakota
  - Gastro Health Research /ID# 164668, Cincinnati, Ohio
  - Duplicate_Duplicate_University Of Cincinnati Medical Center /ID# 164729, Cincinnati, Ohio
  - Cleveland Clinic Main Campus /ID# 209230, Cleveland, Ohio
  - Ohio State University/ Gastroe /ID# 170159, Columbus, Ohio
  - Optimed Research, Ltd. /ID# 205625, Columbus, Ohio
  - Hometown Urgent Care and Resea /ID# 201289, Dayton, Ohio
  - Dayton Gastroenterology, Inc. /ID# 167623, Englewood, Ohio
  - Great Lakes Gastroenterology Research, LLC /ID# 202006, Mentor, Ohio
  - Digestive Disease Specialists /ID# 201063, Oklahoma City, Oklahoma
  - Options Health Research, LLC /ID# 164704, Tulsa, Oklahoma
  - Healthcare Research Consultant /ID# 166244, Tulsa, Oklahoma
  - University of Pennsylvania /ID# 168406, Philadelphia, Pennsylvania
  - Duplicate_Thomas Jefferson University /ID# 168003, Philadelphia, Pennsylvania
  - Pharmacorp Clinical Trials /ID# 165008, Charleston, South Carolina
  - Gastroenterology Associates, P.A. of Greenville /ID# 164643, Greenville, South Carolina
  - Rapid City Medical Center - GI Research /ID# 201733, Rapid City, South Dakota
  - Gastro One /ID# 164730, Cordova, Tennessee
  - Duplicate_East Tennessee Research Institute /ID# 203614, Johnson City, Tennessee
  - Quality Medical Research /ID# 205264, Nashville, Tennessee
  - Vanderbilt University Medical Center /ID# 164607, Nashville, Tennessee
  - TX Clinical Research Institute /ID# 164719, Arlington, Texas
  - Inquest Clinical Research /ID# 164676, Baytown, Texas
  - Texas Digestive Disease Consultants /ID# 209954, Cedar Park, Texas
  - GI Alliance /ID# 209803, Cedar Park, Texas
  - Baylor Scott & White Center for Inflammatory Bowel Diseases /ID# 170161, Dallas, Texas
  - Baylor College of Medicine /ID# 164609, Houston, Texas
  - Centex Studies, Inc. - Houston /ID# 201212, Houston, Texas
  - GI Specialists of Houston /ID# 202340, Houston, Texas
  - Caprock Gastro Research - Lubbock - 80th Street /ID# 215436, Lubbock, Texas
  - Clinical Associates in Research Therapeutics of America, LLC /ID# 164675, San Antonio, Texas
  - Southern Star Research Institute, LLC /ID# 169756, San Antonio, Texas
  - Carl R. Meisner Medical Clinic /ID# 171057, Sugar Land, Texas
  - Tyler Research Institute, LLC /ID# 168679, Tyler, Texas
  - Gastro Health & Nutrition - Victoria /ID# 167810, Victoria, Texas
  - HP Clinical Research /ID# 164631, Bountiful, Utah
  - Advanced Research Institute /ID# 164689, Ogden, Utah
  - Duplicate_Care Access Research /ID# 164685, Salt Lake City, Utah
  - Duplicate_Velocity Clinical Research - Salt Lake City /ID# 166113, West Jordan, Utah
  - Texas Digestive Disease Consultants, PLLC dba GI Alliance /ID# 164728, Bellevue, Washington
  - Virginia Mason Hospital & Medical Center /ID# 164862, Seattle, Washington
  - University of Washington /ID# 164646, Seattle, Washington
  - The Vancouver Clinic, INC. PS /ID# 164874, Vancouver, Washington
  - Froedtert Memorial Lutheran Hospital /ID# 202285, Milwaukee, Wisconsin
  - Allegiance Research Specialists /ID# 165298, Wauwatosa, Wisconsin
- Argentina (6):
  - Cemic /Id# 169183, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Cardio Alem /ID# 211283, San Isidro, Buenos Aires
  - Hospital Italiano de Buenos Aires /ID# 215542, Ciudad Autonoma Buenos Aires, Buenos Aires F.D.
  - Gedyt /ID# 210018, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Hospital Provincial del Centenario /ID# 171251, Rosario, Santa Fe Province
  - Hospital Privado Universitario - Hospital Privado Centro Medico de Cordoba S.A. /ID# 169229, Córdoba
- Australia (6):
  - Concord Repatriation General Hospital /ID# 171506, Concord, New South Wales
  - Coral Sea Clinical Research institute /ID# 212989, North Mackay, Queensland
  - Mater Misericordiae Limited /ID# 204910, South Brisbane, Queensland
  - Royal Adelaide Hospital /ID# 171508, Adelaide, South Australia
  - Box Hill Hospital /ID# 203735, Box Hill, Victoria
  - Fiona Stanley Hospital /ID# 171507, Murdoch, Western Australia
- Austria (3):
  - Klinik Landstrasse /ID# 203438, Vienna, Vienna
  - Medizinische Universitaet Wien /ID# 169459, Vienna, Vienna
  - Landeskrankenhaus Salzburg-Universitaetsklinikum der PMU (LKH) /ID# 214468, Salzburg
- Belgium (5):
  - Cliniques Universitaires UCL Saint-Luc /ID# 200293, Brussels, Brussels Capital
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant /ID# 200295, Yvoir, Namur
  - Duplicate_AZ Sint-Lucas /ID# 200296, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 200031, Leuven, Vlaams-Brabant
  - CHU de Liege /ID# 200294, Liège
- Bosnia and Herzegovina (4):
  - Duplicate_University Clinical Centre of the Republic of Srpska /ID# 200743, Banja Luka, Republika Srpska
  - University Clinical Center Tuzla /ID# 210323, Tuzla, Tuzlanski
  - Clinical Center University of Sarajevo /ID# 201346, Sarajevo
  - Polyclinic and Daily Hospital Dr. Al-Tawil /ID# 217843, Sarajevo
- Brazil (7):
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva /ID# 166853, Goiânia, Goiás
  - Faculdade de Medicina do ABC /ID# 166854, Santo André, La Spezia
  - Hospital Nossa Senhora das Graças /ID# 166856, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre /ID# 166855, Porto Alegre, Rio Grande do Sul
  - Upeclin Fmb - Unesp /Id# 166860, Botucatu, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto /ID# 166859, Ribeirão Preto, São Paulo
  - Kaiser Clinica e Hospital Dia /ID# 166858, São José do Rio Preto, São Paulo
- Bulgaria (3):
  - Duplicate_UMHAT Kaspela EOOD /ID# 167615, Plovdiv
  - Duplicate_Second MHAT Sofia /ID# 167616, Sofia
  - MHAT Trakia /ID# 201677, Stara Zagora
- Canada (17):
  - University of Calgary /ID# 166990, Calgary, Alberta
  - Allen Whey Khye Lim Professional Corporation /ID# 168047, Edmonton, Alberta
  - University of Alberta Hospital /ID# 166987, Edmonton, Alberta
  - Covenant Health /ID# 166996, Edmonton, Alberta
  - Fraser Clinical Trials Inc /ID# 166984, New Westminster, British Columbia
  - Giri Gi Research Institute - Vancouver /ID# 166994, Vancouver, British Columbia
  - QEII - Health Sciences Centre /ID# 169308, Halifax, Nova Scotia
  - Medicor Research Inc /ID# 166997, Greater Sudbury, Ontario
  - London Health Sciences Center- University Hospital /ID# 221039, London, Ontario
  - Scott Shulman Medicine Professional Corporation /ID# 169065, North Bay, Ontario
  - Taunton surgical centre /ID# 168045, Oshawa, Ontario
  - Ottawa Hospital Research Institute /ID# 212412, Ottawa, Ontario
  - Toronto Digestive Disease Associates /ID# 166988, Vaughan, Ontario
  - Hotel Dieu de Levis /ID# 166985, Lévis, Quebec
  - Centre Hospitalier de l'Universite de Montreal - CRCHUM /ID# 170122, Montreal, Quebec
  - Disc_Royal Victoria Hospital / McGill University Health Centre /ID# 170011, Montreal, Quebec
  - CIUSSS de l'Estrie - CHUS /ID# 170936, Sherbrooke, Quebec
- Chile (5):
  - Hospital Guillermo Grant Benavente de Concepción /ID# 212421, Concepción, Bio-Bio
  - CTR Estudios Clinicos /ID# 203940, Providencia, Region Metropolitana Santiago
  - Research Group /ID# 203178, Santiago, Santiago Metropolitan
  - CEC SpA /ID# 169872, Ñuñoa
  - Hospital Clinico Universidad De Los Andes /ID# 207463, Santiago
- China (15):
  - Beijing Friendship Hospital /ID# 204175, Beijing, Beijing Municipality
  - Zhongshan Hospital Xiamen University /ID# 204986, Xiamen, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University /ID# 205227, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University /ID# 204056, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University /ID# 204054, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 204065, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College of HUST /ID# 204051, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University /ID# 204057, Changsha, Hunan
  - Nanjing Drum Tower Hospital /ID# 204899, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 204052, Nanchang, Jiangxi
  - The First Hospital of Jilin University /ID# 206865, Changchun, Jilin
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 204055, Shanghai, Shanghai Municipality
  - The second affiliated hospital of Zhejiang University school of medicine /ID# 204058, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital,Meical School Zhejiang University /ID# 204050, Hangzhou, Zhejiang
  - Duplicate_Tianjin Med Univ General Hosp /ID# 206979, Tianjin
- Colombia (2):
  - Duplicate_Hospital Pablo Tobon Uribe /ID# 202403, Medellín, Antioquia
  - Hospital San Vicente de Paul /ID# 200020, Medellín, Antioquia
- Croatia (6):
  - Clinical Hospital Dubrava /ID# 171165, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Sestre milosrdnice /ID# 171194, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 171168, Zagreb, City of Zagreb
  - Poliklinika Solmed /ID# 211517, Zagreb, City of Zagreb
  - Klinicki Bolnicki Centar KBC Split /ID# 171205, Split, Split-Dalmatia County
  - Zadar General Hospital /ID# 205533, Zadar
- Czechia (4):
  - Nemocnice Ceske Budejovice a.s. /ID# 224390, České Budějovice
  - Hepato-Gastroenterologie HK, s.r.o. /ID# 171564, Hradec Králové
  - ARTROSCAN s.r.o. /ID# 171575, Ostrava
  - ResTrial s.r.o. /ID# 208651, Prague
- Denmark (4):
  - Herlev Hospital /ID# 200785, Herlev, Capital Region
  - Nordsjaellands Hospital /ID# 200788, Hilleroed, Capital Region
  - Kobenhavns Universitet - Hvidovre Hospital (HH) /ID# 200787, Hvidovre, Capital Region
  - Duplicate_Sjaellands Universitets Hospital /ID# 200786, Roskilde, Region Sjælland
- Egypt (7):
  - Alexandria University /ID# 171008, Alexandria, Alexandria Governorate
  - Alexandria University /ID# 171017, Alexandria, Alexandria Governorate
  - National Liver Institute /ID# 170987, Menoufiya, Monufia Governorate
  - Duplicate_Clinical Research Center, Faculty of Medicine, Alexandria university. /ID# 209561, Alexandria
  - National Hepatology and Tropical Medicine Research Institute /ID# 170991, Cairo
  - Ain Shams University Faculty of Medicine /ID# 209566, Cairo
  - Air Force Specialized Hospital /ID# 170993, Cairo
- Estonia (2):
  - West Tallinn Central Hospital /ID# 202787, Tallinn, Harju
  - Tartu University Hospital /ID# 203141, Tartu
- France (16):
  - Chu de Nice-Hopital L'Archet Ii /Id# 171004, Nice, Alpes-Maritimes
  - Duplicate_CHU Bordeaux - Hopital Haut Leveque /ID# 207812, Pessac, Gironde
  - CHU Toulouse - Hopital Rangueil /ID# 169784, Toulouse, Haute-Garonne
  - Duplicate_Hopital Saint Eloi /ID# 170039, Montpellier, Herault
  - Duplicate_CHU Grenoble - Hopital Michallon /ID# 222403, La Tronche, Isere
  - CHRU Nancy - Hopitaux de Brabois /ID# 170970, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHRU Lille - Hopital Claude Huriez /ID# 206653, Lille, Nord
  - CH Valenciennes /ID# 222399, Valenciennes, Nord
  - Centre Hospitalier Universitaire de Saint Etienne - Hopital Nord /ID# 171027, St-Priest-en-Jarez, Pays de la Loire Region
  - HCL - Hopital Lyon Sud /ID# 171030, Pierre-Bénite, Rhone
  - CHU Amiens-Picardie Site Sud /ID# 171023, Amiens, Somme
  - CHRU Tours - Hopital Trousseau /ID# 169783, Chambray-lès-Tours
  - Duplicate_CHU Henri Mondor /ID# 169782, Créteil
  - Clinique Jules Verne /ID# 222240, Nantes
  - Polyclinique Grand Sud /ID# 170037, Nîmes
  - Hopital Beaujon /ID# 171007, Clichy, Île-de-France Region
- Germany (12):
  - Universitatsklinikum Mannheim /ID# 168754, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Ulm /ID# 203554, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen /ID# 203550, Erlangen, Bavaria
  - Duplicate_Agaplesion Markus Krankenhaus /ID# 168753, Frankfurt am Main, Hesse
  - Universitaetsklinikum Frankfurt /ID# 203567, Frankfurt am Main, Hesse
  - Zentrum für Gastroenterologie Saar MVZ GmbH /ID# 206739, Saarbrücken, Saarland
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 168755, Kiel, Schleswig-Holstein
  - Charite Universitaetsklinikum Berlin - Campus Benjamin Franklin /ID# 169271, Berlin
  - Gastroenterologie am Mexikoplatz /ID# 203574, Berlin
  - Universitaetsmedizin Essen St. Josef Krankenhaus Werden /ID# 203569, Essen
  - Universitaetsklinikum Halle (Saale) /ID# 207453, Halle
  - Medizinisches Versorgungszentrum Portal 10 /ID# 200212, Münster
- Greece (6):
  - General Hospital of Athens Ippokratio /ID# 167032, Athens, Attica
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 202102, Athens, Attica
  - Tzaneio general hospital of Piraeus /ID# 206435, Piraeus, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 167031, Heraklion, Crete
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 167033, Athens
  - General Hospital of Thessaloniki Hippokrateio /ID# 208823, Thessaloniki
- Hong Kong (2):
  - Queen Mary Hospital /ID# 171214, Hong Kong
  - Tuen Mun Hospital /ID# 171213, Hong Kong
- Hungary (11):
  - Pecsi Tudomanyegyetem Klinikai Kozpont Mohacsi Korhaz /ID# 209440, Mohács, Baranya
  - CRU Hungary Egeszsegugyi és Szolgaltato Kft. /ID# 205549, Encs, Borsod-Abauj Zemplen county
  - Duplicate_Debreceni Egyetem Klinikai Kozpont /ID# 216420, Debrecen, Hajdú-Bihar
  - Gyongyosi Bugat Pal Korhaz /ID# 201885, Gyöngyös, Heves County
  - Komarom-Esztergom Varmegyei Szent Borbala Korhaz (Clinexpert Tatabanya Kft.) /ID# 209896, Tatabánya, Komárom-Esztergom
  - Kistarcsai Flor Ferenc Korhaz /ID# 206153, Kistarcsa, Pest County
  - Obudai Egeszsegugyi Centrum /ID# 201886, Budapest
  - Duplicate_Semmelweis Egyetem /ID# 210166, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont /ID# 200888, Budapest
  - Debreceni Egyetem Kenezy Gyula Egyetemi Korhaz /ID# 200887, Debrecen
  - Mentahaz Maganorvosi Kozpont /ID# 201888, Székesfehérvár
- Mercy University Hospital /ID# 206512, Cork, Ireland
- Israel (7):
  - Duplicate_Kaplan Medical Center /ID# 170275, Rehovot, Central District
  - Yitzhak Shamir Medical Center /ID# 206449, Ẕerifin, Central District
  - Hadassah Medical Center-Hebrew University /ID# 169926, Jerusalem, Jerusalem
  - Barzilai Medical Center /ID# 223374, Ashkelon, Southern District
  - Soroka University Medical Center /ID# 169911, Beersheba, Southern District
  - Tel Aviv Sourasky Medical Center /ID# 206450, Tel Aviv, Tel Aviv
  - Rabin Medical Center /ID# 202634, Petah Tikva
- Italy (15):
  - Duplicate_IRCCS AOU di Bologna - Policlinico Sant'Orsola-Malpighi /ID# 168155, Bologna, Emilia-Romagna
  - IRCCS Istituto Clinico Humanitas /ID# 168153, Rozzano, Lombardy
  - ASST Fatebenefratelli Sacco - Ospedale Fatebenefratelli e Oftalmico /ID# 168149, Milan, Milano
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 170906, Milan, Milano
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 168156, Rome, Roma
  - Duplicate_Azienda Ospedaliera San Camillo Forlanini /ID# 168152, Rome, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 168150, Rome, Roma
  - Duplicate_IRCCS Ospedale Sacro Cuore Don Calabria /ID# 168154, Negrar, Verona
  - Ospedale Cannizzaro /ID# 168161, Catania
  - Azienda Ospedaliero-Universitaria Renato Dulbecco /ID# 201986, Catanzaro
  - Policlinico San Martino/Univer /ID# 168162, Genova
  - Azienda Ospedaliero-Universitaria di Modena /ID# 200009, Modena
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello /ID# 168157, Palermo
  - Duplicate_Azienda Ospedaliero Universitaria Pisana-Stabilimento di Cisanello /ID# 202419, Pisa
  - Fondazione Policlinico Universitario Campus Bio-Medico /ID# 168151, Roma
- Japan (50):
  - Aichi Medical University Hospital /ID# 165989, Nagakute, Aichi-ken
  - Nagoya University Hospital /ID# 165987, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 165988, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital /ID# 200176, Toyohashi, Aichi-ken
  - National Hospital Organization Hirosaki General Medical Center /ID# 165976, Hirosaki-shi, Aomori
  - Toho University Sakura Medical Center /ID# 165978, Sakura-shi, Chiba
  - Fukuoka University Chikushi Hospital /ID# 214402, Chikushino-shi, Fukuoka
  - Kurume University Hospital /ID# 165996, Kurume-shi, Fukuoka
  - National Hospital Organization Takasaki General Medical Center /ID# 167151, Takasaki-shi, Gunma
  - Duplicate_NHO Fukuyama Medical Center /ID# 167155, Fukuyama-shi, Hiroshima
  - Hiroshima University Hospital /ID# 165998, Hiroshima, Hiroshima
  - Duplicate_Asahikawa Medical University Hospital /ID# 167148, Asahikawa-shi, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 165975, Sapporo, Hokkaido
  - Duplicate_Sapporo Medical University Hospital /ID# 167152, Sapporo, Hokkaido
  - Sapporo IBD Clinic /ID# 223559, Sapporo, Hokkaido
  - Aoyama Clinic /ID# 165993, Kobe, Hyōgo
  - Duplicate_Hyogo Medical University Hospital /ID# 165991, Nishinomiya-shi, Hyōgo
  - Kanazawa University Hospital /ID# 169212, Kanazawa, Ishikawa-ken
  - Iwate Medical University Uchimaru Medical Center /ID# 202465, Morioka, Iwate
  - Imamura General Hospital /ID# 227135, Kagoshima, Kagoshima-ken
  - Idzuro Imamura Hospital /ID# 206655, Kagoshima, Kagoshima-ken
  - Sameshima Hospital /ID# 206677, Kagoshima, Kagoshima-ken
  - Duplicate_Yokohama City University Medical Center /ID# 167156, Yokohama, Kanagawa
  - Japanese Red Cross Kyoto Daiichi Hosital /ID# 165990, Kyoto, Kyoto
  - Duplicate_Kyoto University Hospital /ID# 169887, Kyoto, Kyoto
  - Yokkaichi Hazu Medical Center /ID# 167201, Yokkaichi-shi, Mie-ken
  - Tohoku University Hospital /ID# 167150, Sendai, Miyagi
  - Nara Medical University Hospital /ID# 169213, Kashihara-shi, Nara
  - Kenseikai Dongo Hospital /ID# 208105, Yamatotakada-shi, Nara
  - Duplicate_Niigata University Medical & Dental Hospital /ID# 170042, Niigata, Niigata
  - Ishida Clinic of IBD and Gastroenterology /ID# 167149, Ōita, Oita Prefecture
  - Chikuba Hospital for Proctological and Gastrointestinal Diseases /ID# 165994, Kurashiki-shi, Okayama-ken
  - Duplicate_Okayama University Hospital /ID# 167354, Okayama, Okayama-ken
  - Kinshukai Infusion Clinic /ID# 218873, Osaka, Osaka
  - Osaka Metropolitan University Hospital /ID# 165999, Osaka, Osaka
  - Duplicate_Osaka University Hospital /ID# 169661, Suita-shi, Osaka
  - Osaka Medical and Pharmaceutical University Hospital /ID# 206323, Takatsuki-shi, Osaka
  - Tokitokai Tokito clinic /ID# 165977, Saitama-shi, Saitama
  - Duplicate_Shiga University of Medical Science Hospital /ID# 167157, Ōtsu, Shiga
  - Duplicate_Hamamatsu University Hospital /ID# 224402, Hamamatsu, Shizuoka
  - Duplicate_NHO Shizuoka Medical Center /ID# 167153, Sunto-gun, Shizuoka
  - Institute of Science Tokyo Hospital /ID# 165982, Bunkyo-ku, Tokyo
  - Tokai University Hachioji Hospital /ID# 165984, Hachioji-shi, Tokyo
  - The Jikei University Hospital /ID# 167154, Minato-ku, Tokyo
  - Kyorin University Hospital /ID# 165983, Mitaka-shi, Tokyo
  - Duplicate_Tokyo Women's Medical University Hospital /ID# 205979, Shinjuku-ku, Tokyo
  - Toyama Prefectural Central Hospital /ID# 217836, Toyama, Toyama
  - Japanese Red Cross Wakayama Medical Center /ID# 200641, Wakayama, Wakayama
  - Wakayama Medical University Hospital /ID# 169480, Wakayama, Wakayama
  - Yamagata University Hospital /ID# 200158, Yamagata, Yamagata
- Latvia (3):
  - VCA Polyclinic Aura /ID# 169499, Riga
  - Pauls Stradins Clinical University Hospital /ID# 169494, Riga
  - Duplicate_Digestive Disease Center Gastro /ID# 169518, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 207030, Kaunas
  - Vilnius University Hospital Santaros Klinikos /ID# 203269, Vilnius
- Malaysia (3):
  - Hospital Sultanah Bahiyah /ID# 201317, Alor Star, Kedah
  - Universiti Sains Malaysia /ID# 200101, Kelantan, Kelantan
  - Universiti Kebangsaan Malaysia (UKM) Medical Centre /ID# 170780, Kuala Lumpur, Selangor
- Mexico (3):
  - Instituto de Investigaciones Aplicadas a la Neurociencias A.C. /ID# 207681, Durango, Durango
  - Morales Vargas Centro de Investigacion S.C. /ID# 203496, León, Guanajuato
  - Clinica de Investigacion en Reumatologia y Obesidad S.C. /ID# 206843, Guadalajara, Jalisco
- Netherlands (5):
  - Radboud Universitair Medisch Centrum /ID# 166931, Nijmegen, Gelderland
  - Zuyderland Medisch Centrum /ID# 169699, Heerlen, Limburg
  - Amsterdam UMC, locatie VUmc /ID# 166930, Amsterdam, North Holland
  - Olvg /Id# 166932, Amsterdam, North Holland
  - Medisch Spectrum Twente /ID# 170299, Enschede, Overijssel
- Poland (5):
  - Malopolskie Centrum Kliniczne /ID# 202169, Krakow, Lesser Poland Voivodeship
  - Vistamed /ID# 208571, Wroclaw, Lower Silesian Voivodeship
  - Centrum Zdrowia MDM /ID# 200493, Warsaw, Masovian Voivodeship
  - Duplicate_WIP Warsaw IBD Point Profesor Kierkus /ID# 224302, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Reuma Park /ID# 200489, Warsaw, Masovian Voivodeship
- Portugal (5):
  - Duplicate_Hospital da Senhora da Oliveira Guimaraes, EPE /ID# 170204, Guimarães, Braga District
  - Hospital Egas Moniz /ID# 170232, Lisbon, Porto District
  - Duplicate_Hospital Garcia de Orta, EPE /ID# 170209, Almada, Setúbal District
  - Unidade Local de Saúde do Alto Minho, EPE - Hospital Conde de Bertiandos /ID# 200608, Ponte de Lima, Viana do Castelo District
  - Unidade Local de Saude Sao Joao, EPE /ID# 170211, Porto
- Puerto Rico (2):
  - Mindful Medical Research /ID# 203356, San Juan
  - School of Medicine University of Puerto Rico-Medical Science Campus /ID# 166769, San Juan
- Romania (3):
  - Fundeni Clinical Institute /ID# 167831, Bucharest, București
  - Duplicate_Clinica GASTRO MED SRL /ID# 206363, Cluj-Napoca, Cluj
  - Cabinet Particular Policlinic Algomed /ID# 167832, Timișoara
- Russia (12):
  - Immanuel Kant Baltic Federal University /ID# 203810, Kaliningrad, Kaliningrad Oblast
  - Republican hospital named after V.A. Baranov /ID# 206497, Petrozavodsk, Murmansk Oblast
  - LLC Medical Center /ID# 209234, Novosibirsk, Novosibirsk Oblast
  - Perm Clinical Center of the Federal Medical and Biological Agency /ID# 202989, Perm, Permskiy Kray
  - LLC Novaya Klinika /ID# 206613, Pyatigorsk, Stavropol Kray
  - Professor Pasechnikov Gastroenterology and Pankreatology clinic /ID# 202996, Stavropol, Stavropol Kray
  - Kazan State Medical University /ID# 169589, Kazan', Tatarstan, Respublika
  - Olla-Med Clinic /ID# 208723, Moscow
  - P.A. Bayandin Murmansk Regiona /ID# 169590, Murmansk
  - Euromedservice /ID# 206608, Pushkin
  - X7 Clinical Research Center /ID# 216348, Saint Petersburg
  - City Clinical Hospital No. 31 /ID# 208871, Saint Petersburg
- Serbia (6):
  - Clinical Hosp Center Zvezdara /ID# 168216, Belgrade, Beograd
  - Military Medical Academy /ID# 168785, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 168217, Belgrade, Beograd
  - Clin Hosp Ctr Bezanijska Kosa /ID# 168787, Belgrade, Beograd
  - Duplicate_University Clinical Center Kragujevac /ID# 205856, Kragujevac, Sumadijski Okrug
  - Duplicate_Clinical Center Vojvodina /ID# 168196, Novi Sad, Vojvodina
- Singapore (3):
  - Duplicate_KL Ling Gastroenterology and Liver Clinic /ID# 205739, Singapore, Central Singapore
  - Gleneagles Medical Centre /ID# 206019, Singapore
  - Tan Tock Seng Hospital /ID# 203158, Singapore
- Slovakia (2):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica /ID# 169960, Banská Bystrica, Banská Bystrica Region
  - KM Management, spol. s.r.o. /ID# 170202, Nitra, Nitra Region
- Univ Medical Ctr Ljubljana /ID# 211041, Ljubljana, Slovenia
- South Africa (6):
  - Farmovs (Pty) Ltd /Id# 207534, Bloemfontein, Free State
  - Lenasia Clinical Trial Centre /ID# 205143, Johannesburg, Gauteng
  - Wits Clinical Research /ID# 170850, Johannesburg, Gauteng
  - Allergy & Immunology (AIU) /ID# 171427, Cape Town, Western Cape
  - Dr JP Wright /ID# 170882, Cape Town, Western Cape
  - Private Practice Dr MN Rajabally /ID# 169851, Cape Town, Western Cape
- South Korea (10):
  - Inje University Haeundae Hospital /ID# 202631, Busan, Busan Gwang Yeogsi
  - Dong-A University Medical Center /ID# 167568, Busan, Busan Gwang Yeogsi
  - Duplicate_Pusan National University Hospital /ID# 167565, Busan, Busan Gwang Yeogsi
  - Kyungpook National University Hospital /ID# 207020, Daegu, Daegu Gwang Yeogsi
  - Duplicate_Hanyang University Gurihospital /ID# 167563, Guri-si, Gyeonggido
  - Duplicate_CHA University Bundang Medical Center /ID# 167569, Seongnam-si, Gyeonggido
  - Chungang University Hospital /ID# 207021, Dongjak-gu, Seoul Teugbyeolsi
  - Kangbuk Samsung Hospital /ID# 167562, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 167564, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 167567, Seoul
- Spain (14):
  - Hospital Universitari Son Espases /ID# 201969, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Marques de Valdecilla /ID# 202495, Santander, Cantabria
  - Hospital Universitario Dr. Negrin /ID# 202723, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario de Navarra /ID# 202354, Pamplona, Navarre
  - Duplicate_Hospital Universitario A Coruna - CHUAC /ID# 203909, A Coruña
  - Hospital Universitario Vall d'Hebron /ID# 202721, Barcelona
  - Hospital Clinic de Barcelona /ID# 202726, Barcelona
  - Hospital Universitario de Girona Doctor Josep Trueta /ID# 202644, Girona
  - Hospital Juan Ramon Jimenez /ID# 202727, Huelva
  - Hospital Universitario La Paz /ID# 202725, Madrid
  - Hospital Universitario de Salamanca /ID# 206359, Salamanca
  - Hospital Universitario Virgen Macarena /ID# 202722, Seville
  - Hospital Clinico Universitario de Valencia /ID# 209658, Valencia
  - Hospital Universitario y Politecnico La Fe /ID# 202720, Valencia
- Sweden (6):
  - Hallands Hospital Halmstad /ID# 170815, Halmstad, Halland County
  - Karolinska University Hospital Solna /ID# 224489, Solna, Stockholm County
  - Alingsas lasarett /ID# 170814, Alingsås, Västra Götaland County
  - Sodra Alvsborgs sjukhus /ID# 203078, Borås, Västra Götaland County
  - Duplicate_Sahlgrenska University Hospital /ID# 169032, Gothenburg, Västra Götaland County
  - Duplicate_Sahlgrenska University Hospital /ID# 169170, Gothenburg, Västra Götaland County
- Switzerland (2):
  - Duplicate_Universitatsspital Zurich /ID# 171000, Zurich, Canton of Zurich
  - Inselspital, Universitaetsspital Bern /ID# 170994, Bern
- Taiwan (4):
  - National Taiwan University Hospital /ID# 169805, Taipei City, Taipei
  - China Medical University Hospital /ID# 169803, Taichung
  - Taichung Veterans General Hospital /ID# 169802, Taichung
  - Linkou Chang Gung Memorial Hospital /ID# 169804, Taoyuan
- Turkey (Türkiye) (10):
  - Gazi Universitesi Tip Fakultes /ID# 217445, Yenimahalle, Ankara
  - Acibadem Kozyatagi Hospital /ID# 209404, Kadıköy, Istanbul
  - Sisli Etfal Train & Res Hosp /ID# 171327, Şişli, Istanbul
  - Duplicate_Erciyes University Medical Fac /ID# 171325, Melikgazi, Kayseri
  - Ankara Univ Medical Faculty /ID# 206408, Ankara
  - Inonu Universitesi Turgut Ozal /ID# 201266, Battalgazi/malatya
  - Mustafa Kemal University Medic /ID# 171328, Hatay
  - Duplicate_Istanbul University Istanbul Medical Faculty /ID# 171365, Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi /ID# 171326, Istanbul
  - Mersin University Medical /ID# 171330, Mersin
- Ukraine (6):
  - Lviv Railway Clinical Hospital of branch Healthcare Centers of Public Joint Stoc /ID# 167917, Lviv, Lviv Oblast
  - MNE Vinnytsia Regional Clinical Hospital n.a. M.I.Pyrogov /ID# 222111, Vinnytsia, Vinnytsia Oblast
  - Kharkiv City Clinical Hospital No.2 n.a. Prof. O.O. Shalimov /ID# 167918, Kharkiv
  - Kyiv City Clinical Hospital No.18 /ID# 207890, Kyiv
  - Medical Centre of "Ukrainian German Antiulcer Gastroenterology Centre BYK-KYIV" /ID# 203739, Kyiv
  - MNE KRC Kyiv Regional Clinical Hospital /ID# 202456, Kyiv
- United Kingdom (14):
  - Warrington and Halton Hospitals NHS Foundation Trust /ID# 171396, Warrington, Cheshire West And Chester
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 218830, London, Greater London
  - St George's University Hospitals NHS Foundation Trust /ID# 205550, London, Greater London
  - Taunton and Somerset NHS Foundation Trust /ID# 209666, Taunton, Somerset
  - Mersey and West Lancashire NHS teaching hospitals trust /ID# 209087, Prescot, Warrington
  - Royal United Hospitals Bath /ID# 169062, Bath
  - Ulster Hospital - South Eastern Health & Social Care Trust /ID# 205324, Belfast
  - University Hospitals Birmingham NHS Foundation Trust /ID# 169058, Birmingham
  - The Dudley Group NHS Foundation Trust /ID# 169057, Dudley
  - London North West University Healthcare NHS Trust /ID# 169056, Harrow
  - King's College Hospital NHS Foundation Trust /ID# 169060, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 169063, Newcastle upon Tyne
  - Stockport NHS foundation trust /ID# 208717, Stockport
  - The Royal Wolverhampton NHS Trust /ID# 171395, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Vermeire S, Colombel JF, Danese S, Panaccione R, Peyrin-Biroulet L, Beck K, Chaparro M, Gisbert JP, Dubcenco E, Klaff J, Naling G, Ford S, Remple V, Joshi N, Suravaram S, Duncan B, Wang Y, Wick-Urban B, Loftus EV. Benefit-risk profile of upadacitinib: exploratory post hoc analysis of phase 2b/3 studies in patients with moderately to severely active ulcerative colitis or Crohn's disease. J Crohns Colitis. 2026 Jan 9;20(1):jjaf198. doi: 10.1093/ecco-jcc/jjaf198. PMID 41264726
- [Derived] Dubinsky MC, D'Haens G, Dewit O, Juillerat P, Panaccione R, Fujii T, Dubcenco E, Lacerda AP, Anyanwu SI, Ford S, Cunneen C, Fish I, Joshi N, Garrison A, Loftus EV. Efficacy and Safety with Upadacitinib by Baseline Corticosteroid Use in Patients with Moderately to Severely Active Crohn's Disease. Inflamm Bowel Dis. 2025 Nov 4:izaf250. doi: 10.1093/ibd/izaf250. Online ahead of print. PMID 41189093
- [Derived] Burmester GR, Deodhar A, Irvine AD, Panaccione R, Winthrop KL, Vleugels RA, Levy G, Suravaram S, Palac H, Wegrzyn L, Ford S, Meerwein S, Guttman-Yassky E. Safety Profile of Upadacitinib: Descriptive Analysis in Over 27,000 Patient-Years Across Rheumatoid Arthritis, Psoriatic Arthritis, Axial Spondyloarthritis, Atopic Dermatitis, and Inflammatory Bowel Disease. Adv Ther. 2025 Oct;42(10):5215-5237. doi: 10.1007/s12325-025-03328-y. Epub 2025 Aug 28. PMID 40875187
- [Derived] Panaccione R, Regueiro M, Lee SD, Atreya R, Pedersen G, Broide E, Rodriguez C, van Bodegraven AA, Dubcenco E, Lacerda AP, Feng T, Geng Z, Wang T, van Haaren S, Anyanwu SI, Panes J. Upadacitinib Maintenance Therapy in Crohn's Disease: Final Results From the Randomized Phase 3 U-ENDURE Study. Clin Gastroenterol Hepatol. 2025 Jul 28:S1542-3565(25)00643-3. doi: 10.1016/j.cgh.2025.07.028. Online ahead of print. PMID 40738276
- [Derived] Loftus EV Jr, D'Haens G, Louis E, Regueiro M, Jairath V, Magro F, Nakase H, Dubcenco E, Lacerda AP, Ford S, Feng T, Duncan B, Fish I, Cunneen C, Anyanwu SI, Aponte F, Griffith J, Blumenstein I. Efficacy and safety of upadacitinib maintenance therapy in patients with moderately to severely active Crohn's disease: 2-year results from the U-ENDURE Long-Term Extension study. J Crohns Colitis. 2025 Sep 7;19(8):jjaf138. doi: 10.1093/ecco-jcc/jjaf138. PMID 40704669
- [Derived] Colombel JF, Lacerda AP, Irving PM, Panaccione R, Reinisch W, Rieder F, Steinlauf A, Schwartz D, Feng T, Dubcenco E, Anyanwu SI, Laroux FS, Cunneen C, Powell N. Efficacy and Safety of Upadacitinib for Perianal Fistulizing Crohn's Disease: A Post Hoc Analysis of 3 Phase 3 Trials. Clin Gastroenterol Hepatol. 2025 May;23(6):1019-1029. doi: 10.1016/j.cgh.2024.08.032. Epub 2024 Sep 24. PMID 39326583
- [Derived] Panes J, Louis E, Bossuyt P, Joshi N, Lee WJ, Lacerda AP, Kligys K, Xuan S, Shukla N, Loftus EV Jr. Induction of Endoscopic Response, Remission, and Ulcer-Free Endoscopy With Upadacitinib Is Associated With Improved Clinical Outcomes and Quality of Life in Patients With Crohn's Disease. Inflamm Bowel Dis. 2025 Feb 6;31(2):394-403. doi: 10.1093/ibd/izae200. PMID 39231444
- [Derived] Ghosh S, Feagan BG, Parra RS, Lopes S, Steinlauf A, Kakuta Y, Joshi N, Lee WJ, Lacerda AP, Zhou Q, Xuan S, Kligys K, Shukla N, Louis E. Impact of Upadacitinib Induction and Maintenance Therapy on Health-related Quality of Life, Fatigue, and Work Productivity in Patients with Moderately-to-severely Active Crohn's Disease. J Crohns Colitis. 2024 Nov 4;18(11):1804-1818. doi: 10.1093/ecco-jcc/jjae083. PMID 38835235
- [Derived] Peyrin-Biroulet L, Panaccione R, Louis E, Atreya R, Rubin DT, Lindsay JO, Siffledeen J, Lukin DJ, Wright J, Watanabe K, Ford S, Remple VP, Lacerda AP, Dubcenco E, Garrison A, Zhou Q, Berg S, Anyanwu SI, Schreiber S. Upadacitinib Achieves Clinical and Endoscopic Outcomes in Crohn's Disease Regardless of Prior Biologic Exposure. Clin Gastroenterol Hepatol. 2024 Oct;22(10):2096-2106. doi: 10.1016/j.cgh.2024.02.026. Epub 2024 Mar 15. PMID 38492904
- [Derived] Colombel JF, Hisamatsu T, Atreya R, Bresso F, Thin L, Panaccione R, Parra RS, Ford S, Remple VP, Lacerda AP, Anyanwu SI, Mallick M, Garrison A, Regueiro M. Upadacitinib Reduces Crohn's Disease Symptoms Within the First Week of Induction Therapy. Clin Gastroenterol Hepatol. 2024 Aug;22(8):1668-1677. doi: 10.1016/j.cgh.2024.02.027. Epub 2024 Mar 15. PMID 38492903
- [Derived] Loftus EV Jr, Panes J, Lacerda AP, Peyrin-Biroulet L, D'Haens G, Panaccione R, Reinisch W, Louis E, Chen M, Nakase H, Begun J, Boland BS, Phillips C, Mohamed MF, Liu J, Geng Z, Feng T, Dubcenco E, Colombel JF. Upadacitinib Induction and Maintenance Therapy for Crohn's Disease. N Engl J Med. 2023 May 25;388(21):1966-1980. doi: 10.1056/NEJMoa2212728. PMID 37224198
- See also: Related info — https://www.abbvieclinicaltrials.com/study/?id=M14-430